CLINICAL TRIAL: NCT05245058
Title: A Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of SPH5030 Tablets in Subjects With Advanced Her2-positive Solid Tumors
Brief Title: SPH5030 Tablets in Subjects With Advanced Her2-positive Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPH5030-101
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: HER2-positive Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPH5030 tablets (Experimental): Subjects will take SPH5030 tablets orally on an empty stomach once or twice a day.
  Each subject will receive only one corresponding dose, and there were five dose groups: 50mg/ d, 100mg/ d, 200mg/ d, 300mg/ d and 400mg/ d.
  Interventions: Drug: SPH5030 tablets

INTERVENTIONS:
Drug: SPH5030 tablets — SPH5030 tablets orally once or twice daily.

SUMMARY:
To evaluate the safety and tolerability of SPH5030 tablets in subjects with HER2-positive advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance status of 0 to 1.
2. Life expectancy of more than 3 months.
3. At least one measurable lesion exists.(RECIST 1.1)
4. Histologically or cytologic confirmed HER2 positive metastatic solid tumor which failed prior standard treatment or have no standard treatment.
5. Required laboratory values including following parameters:

   ANC: ≥ 1.5 x 109/L Plt count: ≥ 90x 109/L Hb: ≥ 90 g/L TBIL: ≤ 1.5 x ULN, ALT and AST: ≤ 2.5 x ULN and creatine clearance rate: ULN or≥ 50 mL/min
6. Toxicity from previous antitumor therapy returned to baseline (except for residual hair loss effects) or CTCAE≤ class 1.
7. Blood pregnancy test was negative within 3 days prior to first dose.

Exclusion Criteria:

1. Subjects who have received the prescribed treatment at the prescribed time prior to first dosing.
2. Known active infection within 2 weeks prior to baseline.
3. Subjects with third space fluid that can not be controled.
4. Subjects with uncontrolled or severe cardiovascular disease.
5. Subjects with uncontrolled hypokalemia and hypomagnesemia before study entry.
6. Subjects with severe lung disease.
7. Subjects that are unable to swallow tablets, or dysfunction of gastrointestinal absorption.
8. Using a potent CYP3A4 or CYP2C8 inhibitor or inducer.
9. Steroid treatment for more than 50 days before, or in need of long-term use of steroids.
10. Uncured other tumors within 5 years.
11. Subjects with symptomatic CNS metastasis, pia meningeal metastasis, or spinal cord compression due to metastasis.
12. Evidence of chronic active hepatitis B or C
13. Uncontrolled systemic diseases, including hypertension that cannot be effectively controlled after treatment.
14. Receive any live or attenuated live vaccine within 28 days prior to baseline.
15. Evidence of severe allergies.
16. Evidence of alcohol or drug abuse.
17. Evidence of neurological or psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2025-12-21 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 24 days
  Measurement of DLT of SPH5030 in all subjects
Maximum tolerated dose（MTD） | Up to 24 days
  Measurement of MTD of SPH5030 in all subjects
Number of patients with adverse events | Up to 2 years
  Adverse event type, incidence, duration, correlation with study drug

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of SPH 5030 | Up to 2 years
  To characterize the PK (Pharmacokinetics) of SPH 5030
Time of maximum serum concentration (Tmax) SPH 5030 | Up to 2 years
  To characterize the PK (Pharmacokinetics) of SPH 5030
Area under the serum concentration-time curve (AUC) of the Dosing Interval (0-14) of SPH5030 | Up to 2 years
  To characterize the PK (Pharmacokinetics) of SPH 5030
Area under the serum concentration-time curve (AUC) of the Dosing Interval (0-Last) of SPH5030 | Up to 2 years
  To characterize the PK (Pharmacokinetics) of SPH 5030
Area under the serum concentration-time curve (AUC) of the Dosing Interval (0-infinity) of SPH5030 | Up to 2 years
  To characterize the PK (Pharmacokinetics) of SPH 5030
Accumulation ratio of maximum serum concentration (Rac_Cmax) of SPH5030 | Up to 2 years
  To characterize the PK (Pharmacokinetics) of SPH 5030
Accumulation ratio of area under the serum concentration-time curve (Rac_AUC) of the Dosing Interval (0-14D) of SPH5030 | Up to 2 years
  To characterize the PK (Pharmacokinetics) of SPH 5030
Terminal rate constant(λz) of SPH5030 | Up to 2 years
  To characterize the PK (Pharmacokinetics) of SPH 5030
Half-life (t1/2) of SPH5030 | Up to 2 years
  To characterize the PK (Pharmacokinetics) of SPH 5030
Total clearance(CL) of SPH5030 | Up to 2 years
  To characterize the PK (Pharmacokinetics) of SPH 5030
Volume of distribution(Vz) of SPH5030 | Up to 2 years
  To characterize the PK (Pharmacokinetics) of SPH 5030
Percentage of area under the serum concentration-time curve (AUC) obtained by extrapolation (%AUCex) of SPH5030 | Up to 2 years
  To characterize the PK (Pharmacokinetics) of SPH 5030
Objective Response Rate (Investigator) | Up to 2 years
  Determination of the Objective Response Rate of all patients by investigators
Duration of remission (DOR) | Up to 2 years
  Time from first documentation of objective response (CR or PR) to first documentation of PD/death due to any cause in absence of documented PD, based on central radiology review as per RECIST v1.1.
Disease control rate (DCR) | Up to 2 years
  The proportion of patients with best confirmed RECIST response of CR, PR, or duration of SD.
Progression-free survival (PFS) | Up to 2 years
  The interval between the dates of the first dose of trial treatment until first documentation of disease progression or death, whichever occurs first.
6-month Progression-free Survival (6mPFS) | Up to 2 years
  Number of Patients Achieving 6-month Progression-free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (17):
- China (17):
  - Anhui provincial hospital, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangxi Cancer Hospital, Nanning, Guangxi
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang Cancer Hospital, Anyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Linyi Cancer Hospital, Linyi, Shandong
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu
  - The second people's hospital of neijiang, Neijiang
  - Tianjin Cancer Hospital Airport Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No